CLINICAL TRIAL: NCT06941246
Title: Gingival Crevicular Fluid Levels of Prolactin Hormone in Type 2 Diabetic Patients With Stage III Periodontitis Before and After Non-Surgical Treatments
Brief Title: Prolactin Levels in Type 2 Diabetic Patients With Stage III Periodontitis
Acronym: prolactin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Sara Ibrahim, master's degree student at oral medicine, peridontology ,oral diagnosis and oral Radiology Department, faculty of Dental Medicine for Girls ,Al Azhar university, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-ME-24-04
Record Dates: First submitted 2025-04-12; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus ,Type 2; periodontitis; Gingival Crevicular Fluid; Prolactin; Non- surgical periodontal treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Periodontitis

STUDY DESIGN:
Intervention Model Description: Periodontal Examination At baseline, all participants received a full-mouth clinical examination, and the following periodontal parameters will be recorded: Plaque Index (PI) (19), Gingival Index (GI) (20), Pocket Depth (PD), and Clinical Attachment Loss (CAL).
  Initial periodontal examination, full mouth scaling and root planning (SRP), clinical measurements before and after treatment, gingival crevicular fluid sampling as well as reinforcement of oral hygiene at baseline and during follow-up evaluations will be performed by the same periodontist (E.A.). Reinforcement of oral hygiene will be done every month for 3 months.
  Gingival fluid sampling:
  Gingival crevicular fluid (GCF) collection will be done the second day after clinical examination to prevent the contamination of sample with blood associated with the probing of inflamed sites. Samples will be collected from the buccal aspects of two interproximal sites in teeth that had the highest signs of inflammation and attachment loss
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy (control). (Other): a full-mouth clinical examination, and the following periodontal parameters will be recorded: Plaque Index (PI) (19), Gingival Index (GI) (20), Pocket Depth (PD), and Clinical Attachment Loss (CAL).Gingival fluid sampling: Gingival crevicular fluid (GCF) collection will be done the second day after clinical examination to prevent the contamination of sample with blood associated with the probing of inflamed sites. Samples will be collected from the buccal aspects of two interproximal sites in teeth that had the highest signs of inflammation and attachment loss for periodontitis groups, this will be done before, and 3 months after SRP. For the control group, samples will be collected from the upper first molar.
  The samples will be assayed for PRL by using an enzyme linked immunosorbent assay (ELISA) kits.
  Interventions: Device: paper points; Device: ELISA Kits
- Stage III periodontitis without diabetes (Active Comparator): Periodontal Examination At baseline, all participants received a full-mouth clinical examination, and the following periodontal parameters will be recorded: Plaque Index (PI) (19), Gingival Index (GI) (20), Pocket Depth (PD), and Clinical Attachment Loss (CAL).
  Initial periodontal examination, full mouth scaling and root planning (SRP), clinical measurements before and after treatment, gingival crevicular fluid sampling as well as reinforcement of oral hygiene at baseline and during follow-up evaluations will be performed by the same periodontist (E.A.). Reinforcement of oral hygiene will be done every month for 3 months.
  Gingival fluid sampling:
  Gingival crevicular fluid (GCF) collection will be done the second day after clinical examination to prevent the contamination of sample with blood associated with the probing of inflamed sites.
  Interventions: Procedure: Non Surgical Periodontal Treatment; Device: paper points; Device: ELISA Kits
- Stage III periodontitis with controlled type 2 diabetes (Active Comparator): Periodontal Examination At baseline, all participants received a full-mouth clinical examination, and the following periodontal parameters will be recorded: Plaque Index (PI) (19), Gingival Index (GI) (20), Pocket Depth (PD), and Clinical Attachment Loss (CAL).
  Initial periodontal examination, full mouth scaling and root planning (SRP), clinical measurements before and after treatment, gingival crevicular fluid sampling as well as reinforcement of oral hygiene at baseline and during follow-up evaluations will be performed by the same periodontist (E.A.). Reinforcement of oral hygiene will be done every month for 3 months.
  Gingival fluid sampling:
  Samples will be collected from the buccal aspects of two interproximal sites in teeth that had the highest signs of inflammation and attachment loss
  Interventions: Procedure: Non Surgical Periodontal Treatment; Device: paper points; Device: ELISA Kits
- Stage III periodontitis with uncontrolled type 2 diabetes (Active Comparator): Periodontal Examination At baseline, all participants received a full-mouth clinical examination, and the following periodontal parameters will be recorded: Plaque Index (PI) (19), Gingival Index (GI) (20), Pocket Depth (PD), and Clinical Attachment Loss (CAL).
  Initial periodontal examination, full mouth scaling and root planning (SRP), clinical measurements before and after treatment, gingival crevicular fluid sampling as well as reinforcement of oral hygiene at baseline and during follow-up evaluations will be performed by the same periodontist (E.A.). Reinforcement of oral hygiene will be done every month for 3 months.
  Gingival fluid sampling:
  Samples will be collected from the buccal aspects of two interproximal sites in teeth that had the highest signs of inflammation and attachment loss
  Interventions: Procedure: Non Surgical Periodontal Treatment; Device: paper points; Device: ELISA Kits

INTERVENTIONS:
Procedure: Non Surgical Periodontal Treatment — the intervention includes Non Surgical Periodontal Therapy( scaling and root planning ),performed to reduce periodontal inflammation .Gingival Crevicular fluid samples will be collected before and after treatment to assess changes in prolactin hormone levels.
  Arms: Stage III periodontitis with controlled type 2 diabetes; Stage III periodontitis with uncontrolled type 2 diabetes; Stage III periodontitis without diabetes
Device: paper points — we use paper point to collect GCF sample
Device: ELISA Kits — The samples are analyzed by ELISA kits to measure prolactin levels

SUMMARY:
evaluate the role of prolactin hormone in the pathogenesis of periodontitis by assessing its local gingival levels and assess clinical parameters in patients who have type two diabetes

DETAILED DESCRIPTION:
Periodontal Examination At baseline, all participants received a full-mouth clinical examination, and the following periodontal parameters will be recorded: Plaque Index (PI) (19), Gingival Index (GI) (20), Pocket Depth (PD), and Clinical Attachment Loss (CAL).

Initial periodontal examination, full mouth scaling and root planning (SRP), clinical measurements before and after treatment, gingival crevicular fluid sampling as well as reinforcement of oral hygiene at baseline and during follow-up evaluations will be performed by the same periodontist (E.A.). Reinforcement of oral hygiene will be done every month for 3 months.

Gingival fluid sampling:

Gingival crevicular fluid (GCF) collection will be done the second day after clinical examination to prevent the contamination of sample with blood associated with the probing of inflamed sites. Samples will be collected from the buccal aspects of two interproximal sites in teeth that had the highest signs of inflammation and attachment loss for periodontitis groups, this will be done before, and 3 months after SRP. For the control group, samples will be collected from the upper first molar.

The samples will be assayed for PRL by using an enzyme linked immunosorbent assay (ELISA) kits.

Patient's examinations:

Glycosylated Hemoglobin (Hemoglobin A1c) test and Body Mass Index will be measured to all participants.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 60 years
* Stage III periodontitis
* Type 2 diabetes
* Only patients signing informed written consents

Exclusion Criteria:

* Pregnancy or lactation
* Any known systemic disease
* Any type of previous periodontal treatment (surgical or non-surgical) in the preceding 6 months
* Smoking (former or current)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Prolactin Hormone Levels in Gingival Crevicular Fluid | Baseline and 3 months after non-surgical periodontal treatment
  Gingival crevicular fluid (GCF) will be collected to measure prolactin hormone levels using enzyme-linked immunosorbent assay (ELISA) kits. Samples will be taken from the buccal aspects of two interproximal sites in each participant. Baseline and post-treatment samples will be collected and analyzed. Higher prolactin levels may be associated with more severe inflammation. Unit of Measure :ng/mL

SECONDARY OUTCOMES:
Change in Plaque Index (PI) | Baseline and 3 months after treatment
  The Plaque Index will be measured using the Silness and Löe Index. Scores range from 0 (no plaque) to 3 (abundant plaque on tooth surface). Higher scores indicate worse oral hygiene.reinforcement of oral hygiene at baseline and during follow-up evaluations will be performed by the same periodontist (E.A.). Reinforcement of oral hygiene will be done every month for 3 months. Higher scores indicate worse oral hygiene. Unit of measure: PI Score (0-3)
Change in Gingival Index (GI) | Baseline and 3 months after treatment
  The Gingival Index will be evaluated using the Löe and Silness method. Scores range from 0 (normal gingiva) to 3 (severe inflammation with spontaneous bleeding). Higher scores indicate worse gingival condition. Unit of measure: GI Score (0-3).
Change in Probing Depth (PD) | Baseline and 3 months after treatment
  Probing depth will be measured using a periodontal probe at selected sites. Measurements are recorded in millimeters. Greater probing depth indicates more advanced periodontal destruction. Unit of measure: millimeters (mm)
Change in Clinical Attachment Level (CAL) | Baseline and 3 months after treatment
  Clinical attachment level will be assessed using a periodontal probe to determine the extent of periodontal support loss. Higher values indicate greater tissue damage. Higher values indicate worse periodontal condition Unit of measure: millimeters (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa El wakeel, Professer, Study Director — Al-Azhar University; Zahraa Saeed, lecturer, Study Director — Al-Azhar University; Olfat shaker, profeser, Study Director — Cairo University
Locations (1):
- Sara Ibrahim Hussein Eid, Cairo, Egypt